CLINICAL TRIAL: NCT02808585
Title: Randomized, Double-blind, Placebo-controlled, Multiple-Dose, Study to Assess the Safety, Tolerability, PK and PD After 4 Weeks of Once Weekly Sc. Inj. of PB1046 in Adults With Stable HFrEF, and in Subjects With Cardiac Dysfunction Secondary to DMD
Brief Title: Study to Assess the Safety, Tolerability and PK/PD After 4 Weekly SC Injections of PB1046 in Subjects With Stable HFrEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB1046-PT-CL-0003-P1
Record Dates: First submitted 2016-06-08; First posted 2016-06-22 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — VIP-ELP fusion molecule PB1046

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PB1046 Injection, 0.2 mg/kg (Experimental): Four weekly doses of PB1046 Injection, 0.2 mg/kg
  Interventions: Drug: PB1046 Injection
- PB1046 Injection, 0.4 mg/kg (Experimental): Four weekly doses of PB1046 Injection, 0.4 mg/kg
  Interventions: Drug: PB1046 Injection
- PB1046 Injection, 0.6 mg/kg (Experimental): Four weekly doses of PB1046 Injection, 0.6 mg/kg
  Interventions: Drug: PB1046 Injection
- PB1046 Injection, 1.2 mg/kg (Experimental): Four weekly doses of PB1046 Injection, 1.2 mg/kg
  Interventions: Drug: PB1046 Injection
- Placebo Comparator (Placebo Comparator): Four weekly doses of Placebo (0.9% NaCl) Injection
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: PB1046 Injection — Four weekly subcutaneous injections of PB1046.
  Other Names: PB1046
  Arms: PB1046 Injection, 0.2 mg/kg; PB1046 Injection, 0.4 mg/kg; PB1046 Injection, 0.6 mg/kg; PB1046 Injection, 1.2 mg/kg
Drug: Placebo Injection — Four weekly subcutaneous injections of placebo.
  Other Names: Placebo
  Arms: Placebo Comparator

SUMMARY:
This study will be a sequential multiple-dose escalation study that will enroll (randomize and dose) approximately 28 subjects in four cohorts consisting of 3 active and 1 placebo in Cohort 1 and 6 active and 2 placebo in subsequent cohorts. Randomized subjects will receive a fixed weekly dose of study drug or placebo for a 4 week dosing period.

DETAILED DESCRIPTION:
Qualifying subjects will have a diagnosis of NYHA Class II or III heart failure with a reduced ejection fraction (HFrEF), be in stable condition, and be taking clinician-directed appropriate pharmacological therapy (e.g., angiotensin converting enzyme inhibitors, angiotensin receptor blockers or an evidence based beta blocker) for heart failure at stable doses (with the exception of diuretics) for at least 1 month prior to screening.

During the period between screening and randomization (planned first dose), the study subject will remain on stable pharmacological therapy for heart failure. Also the study subject will be in stable health with no hospitalizations or clinically significant acute illnesses between screening and randomization that would put the subject at increased risk for study participation.

Randomized subjects will receive a fixed weekly dose of study drug or placebo for a 4 week dosing period. Dose escalation in subsequent cohorts will continue if the safety and pharmacokinetic profile are deemed acceptable as assessed by the Study Review Committee.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study-related procedures,
* Male subjects and female subjects of reproductive or childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study drug,
* Body mass index ≥ 18 kg/m2 and ≤ 45 kg/m2,
* Receipt of stable pharmacological therapy(ies) for heart failure for a minimum of 1 month prior to screening and between screening and randomization and are in stable clinical condition,
* NYHA Class II or III heart failure diagnosis (ischemic or non-ischemic confirmed by medical history) at least 6 months prior to screening,
* Stable HF defined as no hospitalizations for cardiac related issues within the previous 3 months prior to the screening visit or between screening and randomization,
* A screening or historical Left Ventricular Ejection Fraction ≤ 40% by centralized reading of 2-D echocardiography,
* Screening hemoglobin ≥ 9.0 g/dL secondary to the volume of blood to be collected during the study period,
* Willing and able to return to the study unit for specified study visits, and be able to self-monitor blood pressure while at home,
* Live and work in an area with reliable cellular services (e.g., Sprint®) for real time transmission of telemetry data to the core laboratory.

Exclusion Criteria:

* Have previously received PB1046 or have a known allergy to the study drug or any of its components,
* Participating in any other study and have received any other investigational medication or device within 30 days prior to screening or are taking part in a non-medication study which, in the opinion of the Investigator, would interfere with study compliance or outcome assessments,
* Diagnosed with acute coronary syndrome (ACS) or an acute myocardial infarction (MI) within 3 months of screening,
* Canadian Cardiovascular Society (CCS) Class III or IV angina necessitating frequent use of as needed short acting nitroglycerin,
* Cardiac surgery or valvuloplasty within 3 months prior to screening,
* Cerebrovascular accident or transient ischemic attack within 3 months prior to screening,
* Sustained systolic blood pressure (SBP) < 110 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg (confirmed by a duplicate seated reading) on at least 3 consecutive readings (self-monitored or office) prior to randomization or overt symptomatic hypotension,
* Sustained resting heart rate >100 beats per minute (BPM) at screening (V1) or prior to randomization,
* History or evidence of clinically significant arrhythmias (uncontrolled by drug therapy or use of an implantable defibrillator), long QT syndrome or evidence of QT prolongation demonstrating QTcF > 460 ms prior to randomization (Subjects with QTcF >460 ms due to electronic pacing by an implanted pacemaker/ICD device may be enrolled),
* Clinically significant renal dysfunction as measured by the estimated glomerular filtration rate (eGFR) of < 40 mL/min/1.73m2 as calculated by the CKD-EPI creatinine-cystatin C equation at screening, or a clinically significant change in renal function between screening and baseline,
* Clinically significant liver dysfunction as measured by: alanine aminotransferase >3.0 × the upper limit of normal (ULN), aspartate aminotransferase >3.0 × the ULN, or serum bilirubin ≥ 1.6 mg/dL at screening, or a clinically significant change in liver function between screening and baseline,
* Pregnant or lactating female subjects,
* Known history of or active alcohol abuse or use of illicit drugs within 1 year prior to randomization,
* Positive screening for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies,
* Any major surgical procedure within 1 month prior to screening or planned surgical procedure during the study period,
* Other medical or psychiatric condition which, in the opinion of the Investigator, would place the subject at increased risk or would preclude obtaining voluntary consent/assent or would confound the secondary objectives of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Phoenix Medical Research, Peoria, Arizona
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - Revivial Research, Miami, Florida
  - North Dallas Research Associates, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Started | 3 | 6 | 7 | 6 | 7
Completed | 3 | 6 | 6 | 4 | 7
Not Completed | 0 | 0 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety/Intent-to-Treat/Per Protocol Population
Groups:
- Total: Total of all reporting groups
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator | Total
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (13.01) | 69.7 (10.89) | 67.6 (11.27) | 64.3 (4.03) | 65 (8.41) | 66.0 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 3 | 2 | 1 | 8
  Male | 1 | 6 | 4 | 4 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 1 | 3
  White | 2 | 5 | 6 | 6 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 7 | 6 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Telemetry
Description: Number of participants with rhythm abnormalities as assessed by continuous mobile telemetry monitoring.
Time Frame: Up to six weeks starting 7 to 10 days before first dose.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
Participants | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: 12-Lead ECG Assessment - Incidence of Clinically Significant Findings
Description: Number of participants with a clinically significant change from baseline in 12-Lead ECG and presence of rhythm abnormalities and relationship to exposure of PB1046 compared to placebo
Time Frame: Seven weeks starting the first week of dosing.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Comparator: Four weekly doses of placebo comparator, 0.9% NaCl.
  PB1046 Injection: Four weekly subcutaneous injections of placebo comparator.
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: 12-Lead ECG - Categorical Analysis of QT/QTc Interval - Participants With Clinically Significant Findings
Description: Number of participants with a clinically significant change from baseline in 12-Lead ECG and presence or absence of rhythm abnormalities and relationship to exposure of PB1046 compared to placebo
Time Frame: Seven weeks starting the first week of dosing.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Laboratory Parameters - Serum Chemistry - Participants With Clinically Significant Findings
Description: Number of participants with clinically significant changes from baseline in laboratory parameters (serum chemistry) and the relationship to PB1046 compared to placebo
Time Frame: Eight weeks starting one week before first dose.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 0 | 1 | 0 | 0 | 0

5. Primary Outcome: Laboratory Parameters - Hematology - Participants With Clinically Significant Findings
Description: Number of participants with clinically significant changes from baseline in laboratory parameters (hematology) and the relationship to PB1046 compared to placebo
Time Frame: Eight weeks starting one week before first dose.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Comparator: Four weekly doses of placebo comparator.
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 1 | 0 | 0 | 0 | 0

6. Primary Outcome: Laboratory Parameters - Urinalysis - Participants With Clinically Significant Findings
Description: Number of participants with clinically significant changes from baseline in laboratory parameters (urinalysis) and the relationship to PB1046 compared to placebo
Time Frame: Eight weeks starting one week before first dose.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Count of Participants; unit: Participants
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 0 | 2 | 0 | 0 | 0

7. Primary Outcome: Laboratory Parameters - eGFR
Description: Changes from baseline in laboratory parameters (eGFR) and the relationship to PB1046 compared to placebo.
  Calculated using Chronic Kidney Disease Epidemiology Collaboration Equation (CKD-EPI)
Time Frame: Baseline, Week 2, 3, 4, 5 and 8.
Population: Safety/Intent-to-Treat/Per Protocol Population. One subject at 0.6 mg/kg dose missed sample collection and was excluded from analysis.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 7
mL/min/1.73m^2
  Week 2 | -1.04 (4.00) | 2.2 (11.41) | -2.9 (13.23) | 1.3 (7.39) | -4.6 (5.88)
  Week 3 | -0.3 (5.77) | 0.2 (10.72) | 2.3 (11.40) | 1.8 (7.57) | -4.6 (5.19)
  Week 4 | 0.0 (2.65) | -1.3 (7.97) | -1.4 (4.12) | 5.8 (9.55) | -6.6 (6.13)
  Week 5 | -0.3 (6.66) | -0.7 (7.26) | -2.2 (13.29) | 9.3 (7.93) | -2.3 (6.63)
  Week 8 | -3.3 (8.62) | -5.7 (11.41) | -3.7 (14.22) | -0.2 (6.79) | -3.0 (4.12)

8. Primary Outcome: Laboratory Parameters - Lipid Profile - Participants With Clinically Significant Findings
Description: Number of participants with clinically significant changes from baseline in laboratory parameters (lipid profile) and the relationship to PB1046 compared to placebo
Time Frame: Eight weeks starting one week before first dose (Baseline and at Week 8).
Measure: Count of Participants; unit: Participants
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Vital Signs - Systolic Blood Pressure
Description: Changes from baseline in vital signs (systolic blood pressure) and the relationship to PB1046 compared to placebo.
Time Frame: Baseline, Day 0, Day 1, 2, 3, 5, 7, 14, 21, 22, 23, 24, 26, 28, 29, 30, 31, and 49.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
mmHg
  Day 0 1 hr | 7.4 (10.88) | -6.2 (19.89) | 3.1 (8.17) | -2.6 (13.43) | 4.6 (17.41)
  Day 0 3 hr | 4.9 (7.17) | -2.6 (14.06) | 1.3 (6.52) | -8.7 (6.24) | 3.4 (11.57)
  Day 1 | -3.4 (2.87) | -5.8 (14.89) | -2.3 (4.79) | -15.4 (18.17) | -7.1 (14.59)
  Day 2 | -0.6 (7.07) | -4.4 (13.45) | -7.2 (7.98) | -8.9 (12.63) | -2.9 (23.54)
  Day 3 | -6.7 (8.25) | 1.8 (24.86) | -8.9 (9.08) | -17.8 (18.09) | -1.8 (16.75)
  Day 5 | 2.4 (11.42) | -4.6 (23.37) | 1.5 (8.57) | -11.7 (20.19) | 1.3 (10.44)
  Day 7 pre | -6.9 (2.22) | -9.4 (11.47) | -5.9 (13.47) | -11.7 (3.78) | -0.3 (10.73)
  Day 14 pre | 4.3 (9.60) | -8.0 (14.73) | -1.6 (9.32) | -8.8 (14.62) | -3.0 (17.71)
  Day 21 pre | -3.0 (6.57) | -8.4 (9.37) | -1.6 (9.32) | -8.8 (14.62) | -5.1 (13.04)
  Day 21 1 hr | -7.9 (4.40) | -14.1 (9.15) | -4.0 (10.00) | -12.8 (15.89) | -3.0 (9.00)
  Day 21 3 hr | -7.9 (4.40) | -14.1 (9.15) | -4.0 (10.00) | -12.8 (15.89) | -3.0 (9.00)
  Day 22 | -5.0 (4.81) | -10.6 (18.27) | -9.4 (10.46) | -20.8 (17.19) | -3.4 (13.67)
  Day 23 | -9.2 (12.16) | -4.7 (9.18) | -9.2 (11.77) | -8.0 (4.33) | -0.8 (11.38)
  Day 24 | 0.9 (5.50) | -1.9 (9.19) | -1.0 (12.16) | -21.6 (29.51) | 2.0 (20.23)
  Day 26 | -8.7 (8.02) | -11.6 (8.41) | -11.4 (5.05) | -9.6 (19.51) | -4.5 (14.75)
  Day 28 | 2.1 (9.83) | -9.4 (13.93) | -8.1 (12.89) | -6.3 (20.28) | -1.2 (21.19)
  Day 29 | 4.2 (12.05) | -7.4 (15.88) | -4.6 (12.30) | -8.9 (7.54) | -3.6 (21.02)
  Day 30 | 0.8 (8.00) | -7.6 (18.85) | -5.9 (9.96) | -11.0 (15.48) | -4.5 (25.36)
  Day 31 | -3.4 (1.35) | -10.4 (17.18) | -9.3 (9.45) | -12.8 (14.83) | -0.2 (13.98)
  Day 49 | 7.1 (14.95) | -6.9 (12.42) | -10.2 (11.97) | -16.8 (22.45) | -3.0 (14.78)

10. Primary Outcome: Vital Signs - Heart Rate
Description: Changes from baseline in vital signs (heart rate) and the relationship to PB1046 compared to placebo.
Time Frame: Baseline, Day 0, Day 1, 2, 3, 5, 7, 14, 21, 22, 23, 24, 26, 28, 29, 30, 31, and 49.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
Beats/min
  Day 0 1 hr | -1.8 (4.55) | -2.1 (6.23) | -2.5 (9.66) | 2.3 (3.64) | -3.0 (5.79)
  Day 0 3 hr | 2.7 (6.49) | -2.4 (5.39) | 0.0 (8.67) | 1.2 (2.83) | 3.0 (9.64)
  Day 1 | -0.7 (1.15) | 4.1 (3.38) | -1.6 (9.66) | 4.1 (5.53) | 3.2 (4.09)
  Day 2 | 1.7 (2.31) | -6.0 (15.58) | -3.3 (8.73) | 2.6 (3.83) | 4.5 (8.66)
  Day 3 | 3.8 (1.35) | -0.8 (5.51) | -2.2 (4.24) | 1.4 (5.86) | -.04 (6.82)
  Day 5 | -1.2 (3.67) | -2.9 (5.06) | -3.2 (9.09) | 2.9 (5.85) | 3.1 (8.62)
  Day 7 pre | 0.6 (2.67) | -0.4 (5.74) | -4.5 (6.05) | 1.6 (1.83) | -1.7 (8.01)
  Day 14 pre | -2.4 (2.14) | -3.7 (6.26) | -0.6 (2.65) | 0.5 (1.29) | -1.9 (7.16)
  Day 21 pre | 3.6 (4.67) | -2.6 (7.62) | -2.7 (2.72) | 0.2 (0.96) | -4.7 (5.84)
  Day 21 1 hr | 3.6 (4.67) | -1.4 (7.49) | 0.9 (2.23) | 1.2 (1.00) | -4.7 (5.84)
  Day 21 3 hr | 8.3 (4.93) | 3.6 (3.62) | -0.9 (3.51) | 0.9 (1.83) | 0.2 (10.92)
  Day 22 | 2.2 (3.02) | -3.3 (10.02) | 0.3 (5.37) | 0.4 (1.07) | 0.3 (8.10)
  Day 23 | -1.8 (1.68) | -2.4 (13.10) | -2.5 (5.92) | 1.4 (1.32) | -0.9 (10.13)
  Day 24 | -2.4 (3.15) | -0.8 (8.52) | -2.1 (4.65) | 1.4 (1.40) | -1.5 (7.49)
  Day 26 | 1.4 (3.91) | -2.2 (10.56) | -1.6 (6.97) | 0.4 (1.13) | -0.8 (7.77)
  Day 28 | -2.0 (8.09) | -0.5 (11.09) | -1.5 (2.10) | 0.2 (1.97) | -2.8 (7.52)
  Day 29 | 0.3 (3.18) | -2.5 (8.62) | -2.1 (9.99) | 2.9 (7.47) | -1.1 (6.84)
  Day 30 | -2.4 (2.50) | -3.9 (11.54) | -3.6 (7.61) | 0.8 (1.67) | 1.7 (8.13)
  Day 31 | -3.4 (3.10) | -4.9 (8.27) | -1.4 (4.96) | -1.6 (1.95) | 0.5 (7.43)
  Day 49 | -2.0 (2.33) | -2.9 (14.19) | -2.3 (4.67) | 1.8 (4.84) | -2.4 (5.70)

11. Primary Outcome: Vital Signs - Temperature
Description: Changes from baseline in vital signs (temperature) and the relationship to PB1046 compared to placebo.
Time Frame: Baseline, Day 0, Day 1, 2, 3, 5, 7, 14, 21, 22, 23, 24, 26, 28, 29, 30, 31, and 49.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
Celsius
  Day 0 1 hr | 0.0 (0.10) | -0.1 (0.35) | 0.0 (0.34) | 0.0 (0.33) | -0.1 (0.28)
  Day 0 3 hr | -0.1 (0.06) | -0.2 (0.36) | 0.0 (0.39) | 0.1 (0.24) | 0.2 (0.53)
  Day 1 | 0.1 (0.12) | -0.3 (0.52) | -0.1 (0.40) | 0.3 (0.14) | 0.2 (0.38)
  Day 2 | -1.1 (2.06) | -0.5 (0.65) | -0.0 (0.45) | 0.1 (0.23) | -0.1 (0.59)
  Day 3 | -1.2 (2.20) | -0.2 (0.46) | 0.0 (0.49) | 0.1 (0.39) | 0.0 (0.66)
  Day 5 | 0.1 (0.21) | -0.2 (0.36) | 0.1 (0.26) | 0.1 (0.39) | 0.0 (0.52)
  Day 7 pre | -0.1 (0.06) | 0.0 (1.22) | 0.1 (0.27) | 0.0 (0.25) | 0.1 (0.37)
  Day 14 pre | -0.2 (0.49) | -0.1 (0.39) | 0.2 (0.27) | 0.1 (0.29) | 0.1 (0.48)
  Day 21 1 hr | 0.1 (0.36) | 0.1 (0.48) | 0.0 (0.42) | 0.1 (0.34) | 0.1 (0.50)
  Day 21 3 hr | 0.1 (0.23) | -0.2 (0.29) | -0.1 (0.39) | -0.1 (0.36) | 0.0 (0.55)
  Day 22 | 0.1 (0.31) | 0.1 (0.24) | 0.2 (0.24) | -0.1 (0.22) | 0.0 (0.49)
  Day 23 | 0.3 (0.25) | 0.2 (0.25) | 0.1 (0.23) | 0.1 (0.26) | 0.1 (0.48)
  Day 24 | 0.3 (0.40) | 0.1 (0.28) | 0.2 (0.30) | -0.1 (0.51) | 0.1 (0.47)
  Day 26 | 0.2 (0.15) | 0.0 (0.66) | 0.1 (0.34) | -0.1 (0.15) | 0.0 (0.44)
  Day 28 | -0.6 (1.42) | 0.2 (0.53) | -0.2 (0.43) | 0.3 (0.30) | 0.0 (0.44)
  Day 29 | 0.1 (0.21) | -0.3 (0.69) | 0.0 (0.40) | 0.1 (0.38) | 0.1 (0.52)
  Day 30 | -1.0 (1.91) | -0.1 (0.69) | 0.1 (0.30) | 0.0 (0.44) | 0.1 (0.51)
  Day 31 | 0.3 (0.25) | 0.1 (0.57) | 0.1 (0.37) | -0.2 (0.29) | -0.1 (0.73)
  Day 49 | 0.1 (0.36) | 0.1 (0.55) | 0.1 (0.42) | 0.0 (0.43) | 8.7 (22.71)

12. Primary Outcome: Vital Signs - Respiratory Rate
Description: Changes from baseline in vital signs (respiratory rate) and the relationship to PB1046 compared to placebo.
Time Frame: Baseline, Day 0, Day 1, 2, 3, 5, 7, 14, 21, 22, 23, 24, 26, 28, 29, 30, 31, and 49.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
Breaths/min
  Day 0 1 hr | 0.7 (1.15) | 0.3 (1.51) | 0.9 (1.57) | -0.3 (1.51) | 0.4 (1.51)
  Day 0 3hr | 1.3 (2.31) | 0.7 (2.07) | 0.0 (1.15) | 0.0 (1.26) | 0.8 (1.83)
  Day 1 | 0.7 (1.15) | 0.3 (2.25) | -0.6 (1.51) | -1.0 (1.10) | 0.3 (1.25)
  Day 2 | 1.0 (1.00) | 0.3 (1.77) | 0.3 (0.76) | -0.3 (1.51) | -0.1 (1.81)
  Day 3 | 0.7 (1.15) | -1.2 (2.15) | 0.3 (2.14) | 0.3 (1.51) | 0.1 (1.07)
  Day 5 | 0.0 (0.00) | 0.4 (1.75) | -0.1 (0.90) | 0.3 (0.082) | 0.6 (1.62)
  Day 21 1hr | -1.3 (1.15) | 0.7 (2.07) | -0.3 (1.51) | -0.5 (1.00) | -0.4 (3.05)
  Day 21 3 hr | 0.0 (2.00) | 0.0 (0.00) | -0.3 (1.97) | 0.5 (1.00) | 0.4 (2.44)
  Day 21 pre | -1.3 (1.15) | 1.0 (3.52) | 0.7 (1.63) | 0.0 (0.00) | 0.6 (1.81)
  Day 22 | 0.0 (2.00) | 1.5 (2.51) | 0.0 (2.19) | -0.5 (1.00) | 0.2 (2.28)
  Day 23 | 0.0 (2.00) | 0.8 (1.60) | -1.0 (2.10) | -0.5 (1.00) | -0.4 (3.15)
  Day 24 | -0.7 (1.15) | 1.2 (2.56) | 0.0 (1.79) | -0.5 (1.00) | 0.2 (1.56)
  Day 26 | -0.7 (1.15) | 1.2 (2.56) | 0.0 (1.79) | -0.5 (1.00) | 0.3 (1.89)
  Day 28 | 0.0 (2.00) | 1.2 (3.37) | 0.3 (1.97) | -0.5 (1.00) | 0.6 (2.44)
  Day 29 | -0.7 (1.15) | 1.7 (3.44) | -0.3 (1.51) | -1.0 (1.15) | -0.3 (2.06)
  Day 30 | 0.7 (1.15) | 1.3 (2.42) | 0.0 (1.26) | -1.0 (1.15) | 0.3 (2.43)
  Day 49 | -0.7 (1.15) | 1.2 (2.40) | 0.7 (1.03) | 0.0 (1.26) | -0.3 (1.38)

13. Primary Outcome: Vital Signs - Diastolic Blood Pressure
Description: Changes from baseline in vital signs (systolic blood pressure) and the relationship to PB1046 compared to placebo.
Time Frame: Baseline, Day 0, Day 1, 2, 3, 5, 7, 14, 21, 22, 23, 24, 26, 28, 29, 30, 31, and 49.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 6 | 4 | 7
mmHg
  Day 0 1 hr | -2.3 (3.38) | -5.7 (13.53) | -2.5 (10.64) | -1.4 (5.68) | 7.8 (9.34)
  Day 0 3 hr | -0.1 (2.50) | -3.1 (11.89) | -4.4 (11.10) | -3.9 (4.08) | 2.6 (3.50)
  Day 1 | -2.7 (1.76) | -1.9 (9.52) | -1.5 (7.77) | -9.5 (11.69) | 3.8 (7.99)
  Day 2 | -0.9 (5.09) | -1.7 (7.48) | -3.0 (9.41) | -5.7 (7.20) | 3.6 (10.18)
  Day 3 | -5.8 (2.17) | 0.1 (10.36) | -2.0 (8.14) | -11.3 (7.33) | 2.8 (7.93)
  Day 5 | 1.1 (7.88) | 1.3 (9.01) | -1.1 (6.61) | -6.9 (12.32) | 1.2 (5.82)
  Day 7 pre | -2.2 (8.60) | -2.5 (6.88) | -1.4 (12.28) | -2.5 (15.60) | 3.6 (6.05)
  Day 14 pre | 3.1 (4.44) | -2.9 (7.07) | -0.2 (7.73) | -4.7 (7.88) | 6.0 (6.28)
  Day 21 pre | 0.7 (2.40) | -1.3 (8.50) | 2.1 (10.83) | -5.8 (5.91) | 4.2 (7.23)
  Day 21 1 hr | -3.4 (1.26) | -4.9 (11.98) | -2.2 (9.70) | -9.8 (6.43) | 2.2 (8.35)
  Day 21 3 hr | -1.4 (3.91) | -7.3 (6.34) | -0.9 (10.82) | -9.8 (8.03) | 4.3 (6.82)
  Day 22 | -2.1 (4.40) | -6.1 (10.52) | -2.2 (9.80) | -10.8 (8.63) | 1.8 (9.89)
  Day 23 | -2.1 (5.00) | -2.1 (8.88) | -3.2 (12.10) | -6.1 (5.39) | 4.5 (7.81)
  Day 24 | 1.0 (2.91) | 1.3 (7.61) | 1.7 (9.05) | -12.8 (14.55) | 3.0 (10.50)
  Day 26 | -1.4 (7.13) | -6.1 (9.86) | -3.2 (10.03) | -6.4 (6.58) | 0.8 (6.74)
  Day 28 | -1.4 (1.58) | -1.4 (9.43) | -0.2 (8.64) | -8.3 (12.66) | 3.7 (10.41)
  Day 29 | 1.6 (7.34) | -2.0 (6.72) | -1.5 (9.98) | -3.7 (9.64) | 2.9 (6.22)
  Day 30 | 2.8 (2.52) | -2.8 (7.92) | -1.9 (11.77) | -8.8 (5.47) | 3.6 (9.02)
  Day 31 | -4.3 (4.04) | -4.6 (10.98) | 0.3 (10.02) | -8.9 (6.10) | 3.9 (6.99)
  Day 49 | 2.6 (2.22) | -3.1 (7.86) | -5.3 (11.08) | -5.0 (10.27) | 5.1 (4.89)

14. Secondary Outcome: Pharmacokinetic Profile - Area Under the Curve Over the Dosing Interval [AUC(0-t)]
Description: Comparison of dose exposures [AUC(0-t)] during once weekly administration of various doses of PB1046
Time Frame: Pre-dose, Day 1 post-dose (1, 3, 24, 48, 72, 120 hours post-dose 1), Day 7, 14, 21 (1, 3, 24, 48, 72, 120 hours post-dose 4), Day 22, 23, 24, 26, 28, 29, 30, and 31.
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: h*ng/mL
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 4
h*ng/mL
  Week 1 | 5791.391 (1639.3) | 12382.716 (4869.3) | 14789.912 (4269.7) | 25555.798 (11248.6)
  Week 4 | 7440.721 (6183.8) | 19007.517 (12655.5) | 16689.657 (7313.0) | 21997.727 (7709.6)

15. Secondary Outcome: Pharmacokinetic Profile - Maximum Serum Concentration (Cmax)
Description: Comparison of dose exposures (Cmax) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 4
ng/mL
  Week 1 | 47.433 (17.3) | 128.317 (64.1) | 218.471 (106.3) | 207.600 (112.3)
  Week 4 | 53.600 (40.2) | 233.450 (189.6) | 211.967 (110.1) | 239.000 (102.6)

16. Secondary Outcome: Pharmacokinetic Profile - Time to Cmax (Tmax)
Description: Comparison of dose exposures (Tmax) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: hours
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 3 | 6 | 6 | 4
hours
  Week 1 | 39.533 (14.1) | 57.594 (54.0) | 27.645 (15.7) | 55.578 (35.8)
  Week 4 | 32.028 (13.7) | 32.042 (12.2) | 36.153 (13.6) | 35.804 (13.9)

17. Secondary Outcome: Pharmacokinetic Profile - Elimination Rate Constant (Lambda z)
Description: Comparison of dose exposures (lambda z) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: 1/hour
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 4
1/hour
  Week 1 | 0.015 (0.0) | 0.018 (0.0) | 0.017 (0.0) | 0.010 (0.0)
  Week 4 | 0.015 (0.0) | 0.026 (0.0) | 0.021 (0.0) | 0.019 (0.0)

18. Secondary Outcome: Pharmacokinetic Profile - Elimination Half-life (t½)
Description: Comparison of dose exposures (t½) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: hours
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 4
hours
  Week 1 | 45.787 (4.7) | 40.806 (7.8) | 54.735 (35.8) | 103.951 (94.6)
  Week 4 | 78.382 (69.3) | 28.333 (6.5) | 34.602 (8.5) | 44.902 (28.5)

19. Secondary Outcome: Pharmacokinetic Profile - Clearance (CL/F), Uncorrected for Bioavailability
Description: Comparison of dose exposures (CL/F) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: mL/h/kg
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 4
mL/h/kg
  Week 1 | 31.992 (10.1) | 33.145 (11.8) | 37.376 (8.2) | 36.067 (15.0)
  Week 4 | 26.981 (16.2) | 28.443 (16.7) | 39.940 (17.7) | 49.220 (11.3)

20. Secondary Outcome: Pharmacokinetic Profile - Volume of Distribution (Vz/F), Uncorrected for Bioavailability (F)
Description: Comparison of dose exposures (Vz/F) during once weekly administration of various doses of PB1046
Time Frame: as for outcome 14
Population: Safety/Intent-to-Treat/Per Protocol Population. Only subjects with sufficient data analyzed.
Measure: Mean (Standard Error); unit: mL/kg
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg
Number analyzed (Participants) | 2 | 6 | 6 | 4
mL/kg
  Week 1 | 2079.049 (451.5) | 1955.795 (826.8) | 2983.922 (1951.6) | 4774.976 (3297.6)
  Week 4 | 3860.362 (4528.5) | 1246.900 (979.1) | 2122.745 (1412.1) | 3401.624 (2650.3)

21. Secondary Outcome: Immunogenicity
Description: Number of participants reporting positive immunogenicity (four-fold increase of pre-dose titer)
Time Frame: Eleven weeks starting the first week of dosing.
Population: Safety/Intent-to-Treat/Per Protocol Population
Measure: Number; unit: subjects
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
Number analyzed (Participants) | 3 | 6 | 7 | 6 | 7
subjects | 2 | 2 | 3 | 6 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | PB1046 Injection, 0.2 mg/kg | PB1046 Injection, 0.4 mg/kg | PB1046 Injection, 0.6 mg/kg | PB1046 Injection, 1.2 mg/kg | Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 0/7 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/7 | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 6/6 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PB1046 Injection, 0.2 mg/kg (N=3) | PB1046 Injection, 0.4 mg/kg (N=6) | PB1046 Injection, 0.6 mg/kg (N=7) | PB1046 Injection, 1.2 mg/kg (N=6) | Placebo Comparator (N=7)
Atrial fibrillation (Cardiac disorders) | NA | 1 | NA | NA | NA
Blood creatinine increased (Cardiac disorders) | NA | 1 | NA | NA | NA
White blood cell count (Cardiac disorders) | NA | 1 | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PB1046 Injection, 0.2 mg/kg (N=3) | PB1046 Injection, 0.4 mg/kg (N=6) | PB1046 Injection, 0.6 mg/kg (N=7) | PB1046 Injection, 1.2 mg/kg (N=6) | Placebo Comparator (N=7)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 3 (20) | 6 (40) | 7 (34) | 6 (28) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (9) | 2 (5) | 2 (10) | 6 (14) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Injection site swelling (General disorders) | 1 (4) | 2 (4) | 4 (5) | 2 (3) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs are not permitted to publish or discuss trial results until 5 years after study completion.

DOCUMENTS (2):
  • Study Protocol (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/85/NCT02808585/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT02808585/SAP_001.pdf